CLINICAL TRIAL: NCT06512675
Title: Effects of an Exercise Program on Reaction Time and Mouse Accuracy in Recreational Video Game Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Timothy Tiu, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20250409
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Quality of Life
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance combined with cardiovascular training group (Experimental): Participants in this group will receive the resistance combined with cardiovascular training intervention for up to 6 weeks
  Interventions: Other: Resistance combined with cardiovascular training

INTERVENTIONS:
Other: Resistance combined with cardiovascular training — Participants will undergo a 6-week exercise program designed under the supervision of a board certified sports medicine physician. The exercise program will consist of a 3 day per week schedule: Monday will be lower body resistance training, Wednesday will be aerobic exercise, and Friday will be upper body resistance training. Each session will be approximately up to 1 hour.

SUMMARY:
This study is intended to evaluate the effects of an exercise program on the change of electronic sports (esports) athletes' reaction time and mouse click accuracy. The benefits of participation are directly related to exercise, and include improved thinking, performance, sleep, and quality of life.

ELIGIBILITY:
Inclusion criteria:

1. Minimum age is 18, and there is no maximum.
2. Must play video games for at least an average of one hour per week
3. University of Miami College student or University of Miami Miller School of Medicine student

Exclusion criteria:

1. Individuals who are not able to participate in a full body exercise program, whether due to injury or an underlying medical condition
2. Individuals who cannot comprehend basic instruction on exercise whether due to a cognitive impairment or language barrier (ie: non English speaker).
3. Conditions that require further medical workup including History or symptoms of cardiac disease, family history of sudden cardiac death, sickle cell disease, history of exercise-related syncope, uncontrolled exercise-associated asthma, acute fractures, active infectious rash, symptoms of relative energy deficiency syndrome, eating disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in participants' physical reaction time | Baseline and up to 6 weeks after starting the program
  Participants' reaction time will be measured in milliseconds using open-source software "Open-source open-access reaction time test"
Change in percentage of participants' mouse click accuracy | Baseline and up to 6 weeks after starting the program
  Participants' mouse click accuracy will be measured as a percentage using a web-based program, "Mouse Accuracy"

SECONDARY OUTCOMES:
Change in participants' number of target efficiency | Baseline and up to 6 weeks after starting the program
  Change in participants' number of target efficiency will be calculated as number of hits divided by possible targets using "Mouse Accuracy"
Change in participants' clicks per second | Baseline and up to 6 weeks after starting the program
  Change in participants' clicks per second will be measured by counting actual mouse clicks per second using "Mouse Accuracy"

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Tiu, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No